CLINICAL TRIAL: NCT07131904
Title: Non-alcoholic, Fiber-enriched Beer and Its Effect on Blood Glucose Concentration: A Scientific Study
Brief Title: Non-alcoholic, Fiber-enriched Beer and Its Effect on Blood Glucose Concentration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Faeh (Other)
Responsible Party: Sponsor-Investigator, David Faeh, Prof. Dr. med. David Fäh, Bern University of Applied Sciences
Organization: Bern University of Applied Sciences (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Fiberbeer trial
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Blood Glucose Concentration; Glycemic Index; Dietary Fiber; Non-alcoholic Beer
Keywords: fiber-enriched beer; functional food; continuous glucose monitoring; postprandial glucose response
MeSH Terms: interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- non-alcoholic, fiber-enriched beer (FEB) (Experimental)
  Interventions: Other: non-alcoholic, fiber-enriched beer (FEB)
- conventional, non-alcoholic beer (Active Comparator)
  Interventions: Other: conventional, non-alcoholic beer
- glucose solution (Active Comparator)
  Interventions: Other: glucose solution

INTERVENTIONS:
Other: non-alcoholic, fiber-enriched beer (FEB) — 500 ml FEB consumed once during a test day in a randomized crossover design. Postprandial blood glucose is monitored for 120 minutes using a continuous glucose monitor (FreeStyle Libre 3).
  Arms: non-alcoholic, fiber-enriched beer (FEB)
Other: conventional, non-alcoholic beer — 500 ml conventional non-alcoholic beer consumed once during a test day in a randomized crossover design. Postprandial blood glucose is monitored for 120 minutes using a continuous glucose monitor (FreeStyle Libre 3).
  Arms: conventional, non-alcoholic beer
Other: glucose solution — Glucose solution containing 12.5 g glucose in 500 ml water, consumed once during a test day in a randomized crossover design. Postprandial blood glucose is monitored for 120 minutes using a continuous glucose monitor (FreeStyle Libre 3).
  Arms: glucose solution

SUMMARY:
This study examines how various non-alcoholic beverages affect blood sugar levels.

The beverages are a non-alcoholic, fiber-enriched beer, a conventional non-alcoholic beer, and a sugar solution. Participants drink one of these beverages on different days. Afterwards, a sensor on the upper arm is used to measure the sugar content in the body fluid under the skin over a period of two hours.

The aim is to find out how much blood sugar concentration rises after drinking. This will be used to check whether the non-alcoholic, fiber-enriched beer has a more favorable effect on sugar metabolism than conventional beverages. Participation is voluntary, and the data will be treated confidentially.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-60 years
* Body mass index (BMI) between 18.5 and 29.9 kg/m²
* Signed informed consent

Exclusion Criteria:

* Diagnosed diabetes
* Gastrointestinal diseases
* Hormonal or other metabolic diseases
* Allergies or intolerances to beer ingredients
* Professional sports (>10 hours/week of intense exercise)
* Special diets (e.g., low-carb, intermittent fasting)
* Sleep disorders or inability to maintain regular sleep (e.g., shift work)
* Pregnancy or breastfeeding
* Smoking
* Inability to speak German or English
* Problems with alcohol, drug, or medication abuse
* Inability to sign informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08-12 (Estimated); Primary Completion 2025-09-22 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Incremental Area Under the Curve (iAUC) for Postprandial Blood Glucose | 0-120 minutes after beverage consumption on each test day
  Incremental area under the curve for interstitial glucose concentration measured over 120 minutes after beverage consumption. Measurements obtained via continuous glucose monitoring (FreeStyle Libre 3) in a randomized crossover design.

SECONDARY OUTCOMES:
Glycemic Index of Fiber-Enriched Beer (FEB) | 0-120 minutes after beverage consumption on each test day
  Glycemic index calculated using the incremental area under the curve for blood glucose after consumption of FEB, compared to glucose solution, according to ISO 26642:2010 methodology.

IPD SHARING:
Plan to Share IPD: Undecided